CLINICAL TRIAL: NCT06644001
Title: Impact of Heyndrickxia (Bacillus) Coagulans Probiotic on Gastrointestinal Function in Healthy Adults: A Randomized Controlled Trial
Brief Title: Bacillus Coagulans Effect on Gastrointestinal Function in Healthy Adults.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kerry Group P.L.C (Industry)
Collaborators: Beijing Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: S23-1464685
Record Dates: First submitted 2024-10-01; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Digestive Discomfort; Constipation; Microbiota
Keywords: GI microbiota, bowel habits, GI symptoms
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Intervention Model Description: A prospective, interventional, randomized, double-blind, parallel, placebo-controlled clinical study. Eligible subjects were randomized at a ratio of 1:1 to receive Bacillus coagulans or placebo once daily for 28 days.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): Bacillus coagulans
  Interventions: Dietary Supplement: Bacillus coagulans GBI-30,6086 (BC GBI-30)
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Bacillus coagulans GBI-30,6086 (BC GBI-30) — 2g powder/sachet, consists of bacillus coagulans at a dose of 1x10^9 CFU, taken once daily before a meal.
  Arms: Probiotic
Dietary Supplement: Placebo — 2g powder/sachet, consists of maltodextrin only, taken once daily before a meal.
  Arms: Placebo

SUMMARY:
A single centre, double-blind, placebo-controlled study to evaluate the effect of the consumption of Bacillus coagulans at a daily dose of 1 x 10⁹ CFU on bowel habits, intestinal microbiota and gastrointestinal symptoms in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

1- Adults male or female aged 18-65 years old. 2- Generally healthy but with irregular bowel movements, including <4 stools/week or periodic (over 2/week) loose stools 2- Agreed not to take other probiotics or prebiotics products during the study period, unless specified by the investigator.

3- Subjects enrolled in the study voluntarily and signed the Consent Form.

Exclusion Criteria:

1. Subjects aged <18 or > 65 years, pregnant or lactating women, and those who are susceptible to allergens or have food allergies.
2. Subjects with cardiovascular, cerebrovascular, hepatic, renal, hematopoietic diseases or endocrine diseases, and or mental illness.
3. Subjects with constipation symptoms caused by surgical operation within the past 30 days; subjects with acute GI track diseases in the past 30 days; subjects with constipation symptoms due to severe organ lesion (colon cancer, severe enteritis, intestinal obstruction, inflammatory bowel disease, etc.)
4. Subjects who could not eat orally or take the study products as prescribed or cannot comply with the protocol.
5. Subjects administered relevant products recently, which would affect the outcome of the study.
6. Subjects who took probiotics or prebiotics products (including yogurt, beverages or foods containing probiotics) within the past month, which may affect the results of the study.
7. Subjects who suffered from gastrointestinal disease within the past month.
8. Subjects who had taken antibiotics in the past month.
9. Subjects who had not taken the test product as prescribed or took other supplements or drugs.
10. Subjects with incomplete data or incomplete information, so that the efficacy could not be estimated.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Stool frequency | 6 weeks period, from enrollment to the end of the study.
  Changes in stool frequency, defined as the number of stools per day. Participants will record their daily stool frequency in a Health Daily Diary. Comparisons will be made between the intervention group and the control group and between timepoints, specifically at each week during the 2-week run-in period and each week from Week 1 to Week 4.
Stool consistency. | 6 weeks period, from enrollment to the end of the study.
  Changes in stool consistency will be assessed using the standard Bristol Stool Scale (BSS). Participants will record their daily stool consistency in a Health Daily Diary. Comparisons will be made between the intervention group and the control group and between timepoints. Specifically, at each week during the 2-week run-in period and each week from Week 1 to Week 4.
Improvement of constipation rate | 6 weeks period, from enrollment to the end of the study.
  Constipation is defined as present if a participant has <4 stools/week and absent if 4 stools/week or more were noted. Analysis will be conducted using data on stool frequency collected by the participants in the Health Daily Diary. Comparisons will be made between groups and between timepoints. Specifically at each week during the 2-week run-in period and each week from Week 1 to Week 4.
Improvement in the defection effort | 6 weeks period, from enrollment to the end of the study.
  Data on symptoms during defection will be collected from the Health Daily Diary and scored as: 0=normal stool habit, 1=defection with mild discomfort, 2= defection with discomfort and difficulty, or 3=defection with frequent abdominal pain or burning. Comparisons will be made between the intervention group and control group and between timepoints. Specifically, at each week during the 2-week run-in period and each week from Week 1 to Week 4.
Changes in intestinal microbiota | 4 weeks period, assessment at Day 0, Day 14 and Day28
  Assessment of changes in the diversity of the fecal microbiota and relative abundance after intervention. Comparisons will be made between groups and between timepoints. Specifically at specifically at baseline (Day 0), Day 14, and Week 28 (end of the study).
Improvement in digestive symptoms scores | 6 weeks; assessment at Day 0, Day 14 and Day 28
  Assessed by the Gastrointestinal Symptom Rates Scale (GSRS).The GSRS has 15 items rated on a seven-point Likert scale from no discomfort to very severe discomfort. These items are grouped into five domains: abdominal pain, reflux, diarrhea, indigestion, and constipation. Scores are the mean of items within each domain, with higher scores indicating more severe symptoms. The overall GSRS score is the average of the five domain scores. Comparisons will be made between the intervention and control groups and at days 0, 14, and 28.
Improvement in upper GI symptoms | 6 weeks; assessment at Day 0, Day 14 and Day 28
  The Severity Of Dyspepsia Assessment (SODA) tool evaluates four symptoms: dyspepsia, heartburn, reflux, and nausea. Each symptom is rated by frequency: 1 (none per week), 2 (once per week), 3 (1-2 times per week), 4 (3-4 times per week), and 5 (daily or more). A decrease in the score over time indicates an improvement in symptoms. Comparisons will be made between the intervention and control groups and at days 0, 14, and 28.

SECONDARY OUTCOMES:
Assessment of the impact of the intervention on the quality of life | 6 weeks; assessment at Day 0, Day 14 and Day 28.
  Changes in Quality of Life (QoL) will be assessed using the 36-Item Short Form Survey (SF-36) version 2. The questionnaire evaluates eight domains of a person's health-related quality of life. Scores for the different domains are converted to a 0-100 scale, where a lower score indicates worse QoL and a higher score reflects better outcome.
Safety assessment-Safety as measured by adverse events | from Day 0 to Day 28
  Documentation of any adverse events to the study product by participants in their daily health diary.
Safety assessment -liver function- Aspartate Aminotransferase (AST) | Day 0 and Day 28
  To assess changes in the Aspartate Aminotransferase blood levels (U/L).
Safety assessment- Liver profile-alanine aminotransferase (ALT) | Day 0 and Day 28
  To assess changes in Alanine Aminotransferase (ALT) blood levels (U/L).
Safety assessment- Liver profile- Bilirubin | Day 0 and Day 28
  To assess changes in blood bilirubin levels (µmol/L).
Safety assessment- Heart rate (vitals) | Day 0, Day 14 and Day 28
  Heart rate (beats per minute)
Safety assessment- Blood pressure (vitals) | Day 0, Day 14 and Day 28
  blood pressure, both of systolic and diastolic (mm Hg)
Safety assessment-ECG findings | Day 0
  Including heart rate (beats per minute), PR Interval (milliseconds), PQ Interval (milliseconds), RR Interval (milliseconds), QRS Interval (milliseconds), and QT Interval (milliseconds), will be recorded.
Safety assessment-urine analysis | Day 0 and Day 28
  To determine any changes in the routine urine analysis test.
Safety assessment-stool analysis | Day 0 and Day 28
  To determine any changes in the routine stool analysis test.
Safety assessment- Chest X-ray findings | Day 0
  Standard Chest X-ray to be checked before the start of the study.
Safety assessment- Kidney profile-Urea | Day 0 and Day 28
  To assess changes in blood urea levels (mmol/L).
Safety assessment- Kidney profile-Creatinine | Day 0 and Day 28
  To assess changes in blood creatinine levels (µmol/L)
Safety assessment- Lipid Profile | Day 0 and Day 28
  To assess changes in blood lipid profile including : Cholesterol (mmol/L), Triglyceride (mmol/L), HDL (mmol/L) and LDL (mmol/L).
Safety assessment- Blood Glucose levels | Day 0 and Day 28
  To assess changes in blood glucose levels (mmol/L)

CONTACTS AND LOCATIONS:
Overall Officials: Gang Hu, MD, Principal Investigator — Beijing Hospital
Locations (1):
- Beijing Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gang H, Wei J, McFarland LV, Zahra R, Saez ME, Blanco-Rojo R, Millette M. Impact of Heyndrickxia (Bacillus) coagulans GBI-30, 6086 (BC30) probiotic on gastrointestinal function in healthy adults: a randomised controlled trial. Benef Microbes. 2025 Jul 22:1-18. doi: 10.1163/18762891-bja00084. Online ahead of print. PMID 40707016